CLINICAL TRIAL: NCT03708120
Title: A Single Group Trial to Determine the Complete Protection Time of an Insect Repellent Formulation Containing 30% Citriodiol® (Oil of Lemon Eucalyptus) Against Three Species of Ticks.
Brief Title: Determining the Complete Protection Time of an Insect Repellent With 30% Citriodiol® Against Three Species of Ticks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCTEC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 593
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Tick Bites
MeSH Terms: conditions — Tick Bites | interventions — Insect Repellents

STUDY DESIGN:
Intervention Model Description: This is a single group trial with the participants acting as their own controls, one arm will be treated with insect repellent, and the other left untreated.
Masking Description: There is no blinding employed since the outcome measures are based on tick behaviour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumer Dose and Tick Repellency (Experimental): Consumer dose: Dosimetry test of insect repellent application to forearms. Tick repellency: Treatment of forearm with insect repellent and exposure to ticks every 15 minutes for 10 hours.
  Interventions: Other: Citrepel (Insect Repellent) EPA Reg. No. 84878-2

INTERVENTIONS:
Other: Citrepel (Insect Repellent) EPA Reg. No. 84878-2 — Citrepel (Insect Repellent) EPA Reg. No. 84878-2 is a pump spray formulation containing the active ingredient Citriodiol®, a tradename for Oil of Lemon Eucalyptus (OLE, Chemical Abstracts Service (CAS) No.: 1245629-80-4). Citriodiol® is derived from Eucalyptus citriodora leaves and contains a minimum of 65% p-Menthane-3,8-diol (PMD, CAS: 42822-86-6) and other constituents occurring naturally in the essential oil source material. The repellent is manufactured by Citrefine International Ltd and will be supplied by them in the pump spray bottle the manufacturer intends to use when the product is marketed with instructions for use on the product label.
  Other Names: Citrapel; Coleman botanicals Insect Repellent

SUMMARY:
This study evaluates the length of time an insect repellent product can protect against three species of ticks. Participants will have one arm treated with the repellent, and throughout the next 10 hours, ticks will be given the opportunity to crawl up the treated arm. The test will stop after 10 hours or when the repellent stops working whichever occurs sooner.

DETAILED DESCRIPTION:
This is a single group trial with the participants acting as their own controls. The study is split into two parts; the first to determine a typical consumer dose when applied to repel ticks, and the second to evaluate the longevity of that consumer dose against three tick species.

To determine the typical consumer dose, twenty-five volunteers will be required to apply the repellent product from final consumer ready pump spray bottle to their forearm. Each volunteer will be asked to read the label and apply the repellent according to the instructions to their forearm. They will repeat the application three times. The amount applied by each subject across the three applications will be averaged, and then the average amount applied by each subject will be averaged to arrive at a "typical consumer dose". This typical consumer dose will be used as the application rate for the tick repellent efficacy trial. Three species are required by the EPA to demonstrate the effectiveness of a repellent. The following tick species have been chosen from the list of five species recommended by the EPA.

Ixodes scapularis - Also known as blacklegged ticks or deer ticks, this species is one of the principal vectors of Lyme disease. They are found in eastern and northern Midwest of the United States. The lifecycle takes approximately two years during which the tick develops from egg to larva, to nymph and finally adult. Larvae, nymphs and adults will all blood feed. Larvae usually feed from smaller mammals and birds, whilst nymphs and adults feed on larger mammals such as deer and humans.

Amblyomma americanum - The Lone Star Tick is found in the eastern United States and in Mexico. This species of hard tick can be a vector of human ehrlichiosis, tularaemia, and may trigger an allergy to the carbohydrate alpha gal found in mammalian meat.

Dermacentor variabilis - The American dog tick is usually found in central and eastern areas of the United States. Adults preferentially feed on large mammals such as dogs and humans, however immature stages will also feed on humans if the opportunity arises. They are the most common vector of Rocky Mountain spotted fever, and can also transmit tularaemia.

Rhipicephalus sanguineus - The brown dog tick is distributed worldwide, including across the United States. It is the vector of many pathogens, including Rickettsia rickettsia, the causative agent of Rocky Mountain spotted fever, Coxiella burnetii, causative agent of Q fever, Ehrlichia canis, and Rickettsia conorii. Dogs are the primary host for the brown dog tick in each of its life stages, but the tick may also bite humans or other mammals.

Ticks will be sourced from disease-free colonies at Oklahoma State University and housed at the London School of Hygiene & Tropical Medicine, United Kingdom, under optimal environmental conditions of 25 ± 3 °C and greater than or equal to 80% Relative Humidity with a 16:8 hour photoperiod.

Single ticks will be exposed to participants' forearms following standardised treatment of one of the participant's forearms with repellent, in a laboratory setting. The treatment will be based on the dose derived from the dosimetry phase of the study, which will be submitted to EPA for review before proceeding to the repellency phase of testing. The treatment will be randomised to either the left or right arm of each participant for each test. There is no blinding employed since the outcome measures are based on tick behaviour. Twenty-five participants will be required for the consumer dose evaluation and to test the repellent against each of the tick species (preferably with a 50:50 ratio of males to females). Participants will test the product at a single dose against at least one of the three species.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with the study procedures
* Able and willing to give fully informed consent
* Male or female
* Aged 18 to 65 years
* Non-smoker or willing to refrain from smoking for 24 hours prior to and during each test
* Able to stand unsupported for periods of at least 5 minutes
* Willing to have hair clipped from the wrist area (3cm upwards from wrist line)

Exclusion Criteria:

* If female, pregnant, nursing or intending to become pregnant, during the time period of the study.
* Not in good general health, including:

  * serious cardiac disorder (whether active or inactive)
  * serious respiratory disorder
  * compromised immune system
  * history of anaphylaxis
* Localised skin disorders affecting the forearms where the product will be applied (including but not restricted to open wounds, eczema, psoriasis, dermatitis or open wounds)
* Participation in another clinical intervention study (excluding biting insect challenge studies*) in the previous 3 months
* Participation in another biting insect challenge study* in the previous 72 hours
* Known or suspected history of tick bite allergies
* Known allergy to Oil of Lemon Eucalyptus, or any ingredients of the test product
* Known phobia of ticks or tick bites
* Employees and spouses of employees of the Study Sponsor (Citrefine Inc.), arctec, and those directly line managed by Professor James Logan
* Students of the Professor James Logan, or any other faculty members involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will report their own gender. The study will aim to enrol approximate equal numbers of males and females.
Enrollment: 70 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
First confirmed crossing | 10 hours
  The time between application of the repellent product and the time at which 1 tick crosses in its entirety into the treated skin and remains there for at least 1 minute, followed within 30 minutes by a second confirmatory crossing.

SECONDARY OUTCOMES:
Average consumer dose | 2 hours
  The mean dose rate applied by a sample of 25 volunteers, measured as mg/cm2 and converted to volume using the specific gravity of the formulation.

CONTACTS AND LOCATIONS:
Overall Officials: James G Logan, Study Chair — ARCTEC
Locations (1):
- ARCTEC, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No